CLINICAL TRIAL: NCT04160351
Title: A Randomised, Open-Label, Cross Over Group, Single-Centre Controlled Study To Evaluate The Clinical Performance Of Medium Cut-Off Membrane Dialyser Compared With High Flux Dialyser In Removing Beta-2- Microglobulin Among Patients With End-Stage Kidney Disease On Chronic Haemodialysis
Brief Title: A Randomised, Open-Label, Cross Over Group, Single-Centre Controlled Study To Evaluate The Clinical Performance Of Medium Cut-Off Membrane Dialyser Compared With High Flux Dialyser Among Patients With Chronic Haemodialysis
Acronym: HD-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selayang Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HS/CTP/HD/001
Record Dates: First submitted 2019-11-05; First posted 2019-11-13 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Hemodialysis-Associated Amyloidosis; Dialysis Amyloidosis; Quality of Life
Keywords: Hemodialysis-Associated Amyloidosis; Dialysis Amyloidosis; Quality of Life

STUDY DESIGN:
Intervention Model Description: This is an open label, cross-over group, single-centre randomised controlled trial comparing MCO Dialyser with High Flux Dialyser in patients with end-stage renal disease on chronic haemodialysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCO Dialyser (Experimental): 12 treatments (4 weeks) with Medium Cut-Off Dialyzer
  Interventions: Device: Theranova 400
- High Flux Dialyser (Active Comparator): 12 treatments (4 weeks) with High Flux Dialyzer
  Interventions: Device: Elisio-19H

INTERVENTIONS:
Device: Theranova 400 — medium cut-off dialyser
  Arms: MCO Dialyser
Device: Elisio-19H — high flux dialyser
  Arms: High Flux Dialyser

SUMMARY:
This is an open label, cross-over group, single-centre randomised controlled trial comparing Medium Cut Off Dialyser with High Flux Dialyser in patients with end-stage renal disease on chronic haemodialysis.

DETAILED DESCRIPTION:
This is an open label, cross-over group, single-centre randomised controlled trial comparing Medium Cut Off(MCO) Dialyser with High Flux Dialyser in patients with end-stage renal disease on chronic haemodialysis.

Patients who are initially on High Flux Dialyser will be randomised into either MCO Dialyser (modality A) or High Flux Dialyser (modality B) dialysate. The dialysate flow (QD) and blood flow (QB) remains unchanged throughout study period. After 12 treatments (4 weeks) a 4-weeks wash-out phase using High-flux dialyzers was performed to minimize carry-over-effects. After the 4-weeks washout phase, the modality is switched to the alternative one for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or above
2. End stage kidney failure receiving hemodialysis for at least 3 years
3. Currently receiving hemodialysis at our center regularly
4. Written informed consent

Exclusion Criteria:

1. Patients with hemodiafiltration
2. Catheter-related blood stream infection in the preceding 4 weeks
3. Malfunctioning of HD catheter
4. Planned transfer to peritoneal dialysis or transplant within 90 days
5. Pregnancy
6. History of active alcohol or substance abuse in the previous 6 months
7. Concurrent participation in another interventional study
8. Other medical condition which, in the investigator's judgment, may be associated with increased risk to the subject or may interfere with study assessments or outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Removal of Beta-2-microglobulin | 4 weeks
  Changes to Beta-2-microglobulin level
Changes to Quality of Life | 27 weeks
  Changes to Quality of life Using SF-36

SECONDARY OUTCOMES:
Inflammatory state after intervention | 4 weeks
  Changes to C-Reactive Protein Level
Changes to Quality of Life | 27 weeks
  Changes to Quality of life Using EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Hin Seng Wong, MD, Study Director — Ministry of Health, Malaysia
Locations (1):
- Selayang Hospital, Batu Caves, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No